CLINICAL TRIAL: NCT03761108
Title: Phase 1/2 FIH Study of REGN5458 (Anti-BCMA x Anti-CD3 Bispecific Antibody) in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Phase 1/2 Study of Linvoseltamab in Adult Patients With Relapsed or Refractory Multiple Myeloma
Acronym: LINKER-MM1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R5458-ONC-1826; 2024-511454-45-00 (EU CTIS Number)
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
Keywords: Relapsed, Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Linvoseltamab - Phase 1 (Experimental): Phase 1 has two parts. Part 1, consists of linvoseltamab intravenous (IV) dose escalation and Part 2, consists of subcutaneous (SC) administration.
  Note: subcutaneous (SC) administration is not applicable for US.
  Interventions: Drug: Linvoseltamab
- Linvoseltamab - Phase 2 - Cohort 1 (Experimental): Low Dose of linvoseltamab IV monotherapy.
  Interventions: Drug: Linvoseltamab
- Linvoseltamab - Phase 2 - Cohort 2 (Experimental): High Dose of linvoseltamab IV monotherapy.
  Interventions: Drug: Linvoseltamab
- Linvoseltamab - Phase 2 - Cohort 3 (Experimental): Anti-interleukin (IL)-6 receptor (R) prophylactic therapy followed by high dose of IV linvoseltamab monotherapy
  Note: Cohort 3 is not applicable for US.
  Interventions: Drug: Linvoseltamab

INTERVENTIONS:
Drug: Linvoseltamab — Administered per the protocol
  Other Names: REGN5458; Lynozyfic™

SUMMARY:
The main purpose of this study is to learn about the safety of linvoseltamab and to find out what is the best dose of linvoseltamab to give to patients with multiple myeloma and to look for any signs that linvoseltamab can effectively treat cancer.

The study is looking at several other research questions, including:

* Side effects that may be experienced by people receiving linvoseltamab
* How linvoseltamab works in the body
* How much linvoseltamab is present in the blood
* How linvoseltamab may work to treat cancer

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
2. Confirmed diagnosis of active Multiple Myeloma (MM) by International Myeloma Working Group (IMWG) diagnostic criteria
3. Patients must have myeloma that is response-evaluable according to the 2016 IMWG response criteria as defined in the protocol.

   * Phase 1, Part 1 (Dose Escalation): Patients with MM who have exhausted all therapeutic options that are expected to provide meaningful clinical benefit, either through disease relapse, treatment refractory disease or intolerance of the therapy and including either:

     a. Progression on or after at least 3 lines of therapy, or intolerance of therapy, including a proteasome inhibitor, an Immunomodulatory agent (IMiD), and an anti-CD38 antibody, OR b. Progression on or after an anti-CD38 antibody and have disease that is "double refractory" to a proteasome inhibitor and an IMiD, or intolerance of therapy. The anti-CD38 antibody may have been administered alone or in combination with another agent such as a proteasome inhibitor (PI). Refractory disease is defined as lack of response or relapse within 60 days of last treatment.
   * Phase 1, Part 2 (SC Administration): Patients with MM whose disease meets the following criteria:

     a. Progression on or after at least 3 prior lines of therapy including a(n) PI, IMiD, and anti-CD38 antibody, OR b. Patients must be triple-refractory, defined as being refractory to prior treatment with at least 1 anti-CD38 antibody, a proteasome inhibitor, and an IMiD.
   * Phase 2 (Cohorts 1 and 2):

   Patients with MM whose disease meets the following criteria:

   a. Progression on or after at least 3 prior lines of therapy including a(n) PI, IMiD, and anti-CD38 antibody, OR b. Patients must be triple- refractory, defined as being refractory* to prior treatment with at least 1 PI, 1 IMiD, and an anti-CD38 antibody.
   * Phase 2 (Cohort 3):

   Patients with MM whose disease meets the following criteria:
   1. Progression on or after at least 3 prior lines of therapy including a(n) PI, IMiD, and anti-CD38 antibody, OR
   2. Patients must be triple- refractory, defined as being refractory* to prior treatment with at least 1 PI, 1 IMiD, and an anti-CD38 antibody.

      * Refractory disease is defined as progression during treatment or within 60 days after completion of therapy, or <25% response to therapy.

   AND, for ALL patients, if they have relapsed after a BCMA-directed CAR-T cellular therapy then:

   • Treatment with a CAR-T must have been associated with a response of PR or better, and

   • If CAR-T cellular therapy was the most recent prior therapy, excluding corticosteroids, then treatment must have been a minimum of 60 days prior to treatment with linvoseltamab.

   Key Exclusion Criteria:

1. Diagnosis of plasma cell leukemia, primary systemic light-chain amyloidosis, (excluding myeloma-associated amyloidosis), Waldenström macroglobulinemia (lymphoplasmacytic lymphoma), or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) 2. Patients with known MM brain lesions or meningeal involvement 3. Cardiac ejection fraction <40% by echocardiogram or multi-gated acquisition scan (MUGA) 4. Prior treatment with BCMA-directed immunotherapies, including BCMA bispecific antibodies and BiTEs. Note: BCMA antibody-drug conjugates are not excluded and BCMA-directed CAR-T treatment is not excluded in Phase 2 Cohort 3.

5. History of allogeneic stem cell transplantation at any time, or autologous stem cell transplantation within 12 weeks of the start of study treatment

Note 1: Other protocol defined inclusion / exclusion criteria apply Note 2: US sites are active but currently not enrolling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2033-03-30 (Estimated); Study Completion 2033-06-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) from the first dose through the end of the DLT observation period | Up to 28 days
  Phase 1 and Phase 2 for Japanese cohort only
Incidence and severity of treatment-emergent adverse events (TEAEs) | Up to 5 years
  Phase 1 Note: Phase 1, part 2 is not applicable for US.
Incidence and severity of adverse events of special interest (AESI) | Up to 5 years
  Phase 1 Note: Phase 1, part 2 is not applicable for US.
Assessment of the pharmacokinetics (PK) of linvoseltamab | Up to 5 years
  Phase 1 part 2 Note: Phase 1, part 2 is not applicable for US.
Concentrations of linvoseltamab in serum over time | Up to 5 years
  Phase 2, for Japanese cohort only
Objective response rate (ORR) as determined by an Independent Review Committee (IRC) | Up to 5 years
  Phase 2, cohorts 1 and 2
Incidence and severity of cytokine release syndrome (CRS) with linvoseltamab | Up to 5 years
  Phase 2, cohort 3 Note: Phase 2, Cohort 3 is not applicable for US.
ORR of IV linvoseltamab as assessed by investigator | Up to 5 years
  Phase 2, cohort 3 Note: Phase 2, Cohort 3 is not applicable for US.

SECONDARY OUTCOMES:
Concentrations of linvoseltamab in the serum over time | Up to 5 years
  Phase 1 part 1 and Phase 2 Note: Phase 2, Cohort 3 is not applicable for US.
Incidence over time of anti-drug antibodies (ADAs) to linvoseltamab | Up to 5 years
  Phase 1 and Phase 2 Note: Phase 1, part 2 and Phase 2, Cohort 3 is not applicable for US.
Titer of anti-drug antibodies (ADAs) to linvoseltamab over time | Up to 5 years
  Phase 1 and Phase 2 Note: Phase 1, part 2 and Phase 2, Cohort 3 is not applicable for US.
Incidence of neutralizing antibodies (NAb) to linvoseltamab over time | Up to 5 years
  Phase 1 and Phase 2 Note: Phase 1, part 2 and Phase 2, Cohort 3 is not applicable for US.
Duration of response (DOR) as determined by an IRC, measured using the IMWG criteria | Up to 5 years
  Phase 2, cohorts 1 and 2
DOR as determined by an investigator, measured using the International Myeloma Working Group (IMWG) criteria | Up to 5 years
  Phase 1 and Phase 2 Note: Phase 1, part 2 is not applicable for US.
Progression-free survival (PFS) as determined by an IRC, measured using the IMWG criteria | Up to 5 years
  Phase 2
PFS as determined by an investigator, measured using the IMWG criteria | Up to 5 years
  Phase 1 and Phase 2 Note: Phase 1, part 2 is not applicable for US.
Rate of minimal residual disease (MRD) negative status, using the IMWG criteria | Up to 5 years
  Phase 1 Note: Phase 1, part 2 is not applicable for US.
Rate of MRD negative status | Up to 5 years
  Phase 2 Note: Phase 2, Cohort 3 is not applicable for US.
Overall survival (OS) | Up to 5 years
  Phase 1 and Phase 2 Note: Phase 1, part 2 and Phase 2, Cohort 3 is not applicable for US.
ORR as measured as determined by blinded IRC, as measured using the IMWG criteria | Up to 5 years
  Phase 1, part 1 dose level 7 (DL7)
ORR as determined by the investigator, measured using the IMWG criteria | Up to 5 years
  Phase 1 and Phase 2 Note: Phase 1, part 2 is not applicable for US.
Effects of linvoseltamab on health-related quality of life (HRQoL) and patient-reported symptoms and functioning per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) | Up to 5 years
  Phase 2
  The EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including global health status/quality of life, functional Scales (physical, role, emotional, cognitive, and social), symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Participants rate items on a 4-point scale, with 1 as "not at all" and 4 as "very much."
  Note: Phase 2, Cohort 3 is not applicable for US.
Effects of linvoseltamab on HRQOL and patient-reported symptoms and functioning per Quality of Life Questionnaire-Multiple Myeloma module 20 [QLQ-MY20]) | Up to 5 years
  Phase 2
  The EORTC QLQ-MY20 is a self -administered instrument to assess QoL in persons with MM. This 20-item questionnaire measures the following domains: symptom scales, including disease symptoms (6 items) and symptoms related to side effects of treatment (10 items); function scale and future perspective (3 items); and body image (1 item). A high score represents a high level of symptoms or problems.
  Note: Phase 2, Cohort 3 is not applicable for US.
Effects of linvoseltamab on HRQOL and patient-reported symptoms and functioning per EuroQoL-5 Dimension-3 Level Scale [EQ-5D-3L]) | Up to 5 years
  Phase 2
  The EQ-5D-3L is a self-administered generic standardized health status measure, consisting of an EQ-5D descriptive system and an EQ visual analog scale. The EQ-5D-3L descriptive system assesses 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 3-level scale: no problems, some problems, and extreme problems. The EQ visual analog scale component is a vertical visual analog scale used by patients to rate their health.
  Note: Phase 2, Cohort 3 is not applicable for US.
Change in patient-reported global health status/QoL per EORTC QLQ-C30 | Baseline up to Up to 5 years
  Phase 2 Note: Phase 2, Cohort 3 is not applicable for US.
Time to definitive deterioration in patient-reported global health status/QoL per EORTC QLQ-C30 | Up to 5 years
  Phase 2 Note: Phase 2, Cohort 3 is not applicable for US.
Effects of linvoseltamab on general health status per EQ-5D-3L | Up to 5 years
  Phase 2 Note: Phase 2, Cohort 3 is not applicable for US.
Effects of linvoseltamab on patient-reported functions and symptoms per EORTC QLQ-C30 | Up to 5 years
  Phase 2 Note: Phase 2, Cohort 3 is not applicable for US.
Effects of linvoseltamab on patient-reported functions and symptoms per QLQ-MY20 | Up to 5 years
  Phase 2 Note: Phase 2, Cohort 3 is not applicable for US.
Incidence and severity of TEAEs with linvoseltamab | Up to 5 years
  Phase 2 Note: Phase 2, Cohort 3 is not applicable for US.
Incidence and severity of AESIs with linvoseltamab | Up to 5 years
  Phase 2 Note: Phase 2, Cohort 3 is not applicable for US.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (40):
- United States (14):
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center - McKinley Drive, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Indiana University_Michigan Street, Indianapolis, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - C. S. Mott_University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Ohio State University James Cancer Hospital, Columbus, Ohio
  - Oregon Health and Science University (OHSU) Marquam Hill Campus, Portland, Oregon
  - University of Texas MD Anderson Clinic, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
- Belgium (2):
  - ZNA Psychiatrisch Ziekenhuis Stuivenberg, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
- Germany (3):
  - Universitatsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg Universitaet Mainz KoeR, Mainz, Rhineland-Palatinate
  - Universitatsklinikum Wurzburg, Würzburg
- Japan (10):
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Gunma University Hospital, Maebashi, Gunma
  - Ibaraki Prefectural Central Hospital, Kasama-shi, Ibaraki
  - University Hospital Kyoto Prefectural Univ of Medicine, Kyoto, Kyoto
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Tokushima Prefectural Central Hospital, Tokushima, Tokushima
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - Keio University Hospital, Tokyo
- South Korea (4):
  - Center for Hematologic Malignancy, Goyang-si, Gyeonggi-do
  - Seoul National University Cancer Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Yonsei University College of Medicine, Severance Hospital, Seoul
- Spain (6):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Universitary Hospital La Princesa, Madrid, Salamanca
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
- Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers may request access to study documents (including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan) that support the methods and findings reported in a manuscript. Individual de-identified participant data will be made available once the indication has been approved by a regulatory body, if there is participant consent and there is not a reasonable likelihood of participant re-identification.
URL: https://vivli.org/

REFERENCES:
- [Derived] Lee HC, Zonder JA, Dhodapkar MV, Jagannath S, Hoffman JE, Suvannasankha A, Shah MR, Lentzsch S, Baz R, Maly JJ, Namburi S, Pianko MJ, Ye JC, Wu KL, Silbermann R, Min CK, Vekemans MC, Munder M, Byun JM, Martinez-Lopez J, DeVeaux M, Roccia T, Chokshi D, Seraphin M, Knorr K, Boyapati A, Hazra A, Rodriguez Lorenc K, Kroog GS, Bumma N, Richter J. Linvoseltamab in Patients With Relapsed/Refractory Multiple Myeloma in the LINKER-MM1 Study: Longer Follow-Up and Subgroup Analyses. Clin Lymphoma Myeloma Leuk. 2025 Nov 12:S2152-2650(25)04283-1. doi: 10.1016/j.clml.2025.11.004. Online ahead of print. PMID 41387038
- [Derived] Bumma N, Richter J, Jagannath S, Lee HC, Hoffman JE, Suvannasankha A, Zonder JA, Shah MR, Lentzsch S, Baz R, Maly JJ, Namburi S, Pianko MJ, Ye JC, Wu KL, Silbermann R, Min CK, Vekemans MC, Munder M, Byun JM, Martinez-Lopez J, Cassady K, DeVeaux M, Chokshi D, Boyapati A, Hazra A, Yancopoulos GD, Sirulnik LA, Rodriguez Lorenc K, Kroog GS, Houvras Y, Dhodapkar MV. Linvoseltamab for Treatment of Relapsed/Refractory Multiple Myeloma. J Clin Oncol. 2024 Aug 1;42(22):2702-2712. doi: 10.1200/JCO.24.01008. Epub 2024 Jun 16. PMID 38879802